CLINICAL TRIAL: NCT06371677
Title: Polish Nationwide Register of Hospitalized Patients in Cardiac Intensive Care Units
Acronym: POL-CICU
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: KB/2024
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Shock; Death; Cardiac Intensive Care Unit; Treatment Complication; Stroke; Multiple Organ Failure; Infections
MeSH Terms: conditions — Shock; Death; Stroke; Multiple Organ Failure; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac Intensive Care Units (CICUs) provide care for a diverse patient population. Understanding the clinical characteristics, analysis of treatment modalities, and prognosis of patients hospitalized in the CICU are important to improve cardiovascular care. The purpose of this registry is to determine the demographics, clinical, treatment, and prognosis of patients hospitalized in the Polish CICUs. Data from this multicenter, prospective observational study will provide more robust data to facilitate quantitative characterization of cardiac care in contemporary Polish CICUs and enable the development of infrastructure for clinical trials in CICUs.

ELIGIBILITY:
All consecutive patients hospitalized at Polish CICUs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All consecutive patients hospitalized at Polish CICUs.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 01.10.2024 - 31.03.2025

SECONDARY OUTCOMES:
Shock (cardiogenic/hypovolemic/anaphylactic/septic/neurogenic/obstructive) | 01.10.2024 - 31.03.2025
Treatment-related complications (tamponade, dissection, stroke, embolism, etc.) | 01.10.2024 - 31.03.2025

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kowalik, MD, PhD, Principal Investigator — 1st Department of Cardiology, Medical University of Warsaw; Monika Gawałko, MD, PhD, Principal Investigator — 1st Department of Cardiology, Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: Undecided